CLINICAL TRIAL: NCT04469829
Title: Methotrexate Versus Secukinumab Safety in Psoriasis Patients With Metabolic Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Paolo Gisondi, Prof, Universita di Verona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gisondi5
Record Dates: First submitted 2020-07-02; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Psoriasis; Metabolic Syndrome
Keywords: psoriasis; methotrexate; secukinumab; metabolic syndrome; safety
MeSH Terms: conditions — Psoriasis; Metabolic Syndrome | interventions — secukinumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- secukinumab (Experimental): patients with psoriasis and metabolic syndrome candidate for treatment with secukinumab standard doses
  Interventions: Drug: Secukinumab
- methotrexate (Active Comparator): patients with psoriasis and metabolic syndrome candidate for treatment with methotrexate dosed 15 mg/week
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Secukinumab — standard doses of secukinumab for psoriasis
  Arms: secukinumab
Drug: Methotrexate — Methotrexate 15 mg/week
  Arms: methotrexate

SUMMARY:
A prospective, controlled, open trial in psoriasis patients with metabolic syndrome, candidate to methotrexate or secukinumab was conducted between January 2019 and May 2020. The primary end point of the study was investigating any variations in waist circumference, body mass index (BMI), blood pressure, fasting glucose, total cholesterol, low density lipoprotein (LDL)-cholesterol, high density lipoprotein (HDL)-cholesterol, triglycerides, aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatinine levels between baseline and month-6 and 12 of follow-up.

DETAILED DESCRIPTION:
A prospective, non-randomized controlled open trial in psoriasis patients with metabolic syndrome was conducted between January 2019 and May 2020. Inclusion criteria were age ≥ 18 years, being affected by moderate to severe chronic plaque psoriasis and concomitant metabolic syndrome and being candidate to systemic treatment with methotrexate or secukinumab according to the Italian guideline for psoriasis. Psoriasis was diagnosed on clinical base, and it was classified as moderate to severe if PASI ≥ 10, Investigator Global Assessment (IGA) score≥ 3 and/or Dermatology Life Quality Index ≥ 10%. Metabolic syndrome was diagnosed according to criteria of the National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III) and The American Heart Association and the National Heart, Lung, and Blood Institute (AHA/NHLB).3 In particular, metabolic syndrome was confirmed in presence of at least three of the following components: abdominal obesity (waist circumference ≥ 102 cm for men or ≥ 88 cm for women), triglycerides ≥ 150 mg/dL, HDL cholesterol ≤ 40 mg/dL for men or 50 mg/dL for women, systolic/diastolic blood pressure ≥ 130/85 mmHg or receiving drug treatment, and fasting plasma glucose ≥ 100 mg/dL. Exclusion criteria were being affected by psoriatic arthritis, pregnancy, breast feeding, having initiated a systemic treatment for psoriasis in the previous 3 months and having a clinical condition that could affect the metabolic parameters other than metabolic syndrome. After having signed the informed consent for the participation in the study, eligible patients were consecutively assigned in a 1:1 ratio to secukinumab (standard dose) or methotrexate 15 mg/week by subcutaneous administration and folic acid supplementation 5 mg given 24 hours after methotrexate. The primary endpoint was investigating any variation in waist circumference, body mass index (BMI), blood pressure, fasting glucose, total cholesterol, low density lipoprotein (LDL)-cholesterol, high density lipoprotein (HDL)-cholesterol, triglycerides, aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatinine levels at month-6. Any other adverse events related to the treatments and the proportion of patients who discontinued the treatment because of adverse reactions were also reported. The secondary endpoints were assessing the PASI 75 and PASI 90 proportion of responders in the two groups at 6 and 12 months follow-up. Clinical and laboratory data were evaluated at the baseline and every 3 months up to month 12.

Statistical Methods A descriptive statistic was conducted using proportions for categorical and mean and standard deviation (SD) for quantitative variables. The categorical variables were compared between the groups using the chi-squared test, while the quantitative variables were compared using the Student's T test. Variations in waist circumference, BMI, blood pressure, fasting glucose, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, AST, ALT, creatinine levels between baseline and month-6 or 12 were assessed by paired t-test in patient receiving methotrexate or secukinumab, respectively. PASI 75 and PASI 90 proportion of responders at month -6 or 12 in the two cohorts' were compared by the chi-squared test. The normal distribution of data was confirmed using the one-sample Kolmogorov-Smirnov Test. A value of p< 0.05 was considered statistically significant. Statistical analysis was performed using the STATA (version 13 StataCorp, College Station, TX, U.S.A.).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* being affected by moderate to severe chronic plaque psoriasis and concomitant metabolic syndrome
* being candidate to systemic treatment with methotrexate or secukinumab according to the Italian guideline for psoriasis

Exclusion Criteria:

* being affected by psoriatic arthritis, pregnancy, breast feeding,
* having initiated a systemic treatment for psoriasis in the previous 3 months and having a clinical condition that could affect the metabolic parameters other than metabolic syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in waist circumference at month 12 | 12 month
  Changes in waist circumference at month 12
Changes in BMI at month 12 | 12 month
  Changes in BMI at month 12
Changes in blood pressure at month 12 | 12 month
  Changes in blood pressure at month 12
Changes in fasting glucose at month 12 | 12 month
  Changes in fasting glucose at month 12
Changes in total cholesterol at month 12 | 12 month
  Changes in total cholesterol at month 12
Changes in LDL cholesterol at month 12 | 12 month
  Changes in LDL cholesterol at month 12
changes in (HDL)-cholesterol at month 12 | 12 month
  changes in (HDL)-cholesterol at month 12
Changes in triglycerides at month 12 | 12 month
  Changes in triglycerides at month 12
Changes in AST at month 12 | month 12
  Changes in AST at month 12
Changes in ALT at month 12 | month 12
  Changes in ALT at month 12

SECONDARY OUTCOMES:
PASI75 and PASI90 | 6 and 12 months
  assessing the PASI 75 and PASI 90 proportion of responders in the two groups at 6 and 12 months follow-up

OTHER OUTCOMES:
adverse reactions | 6 and 12 months
  other adverse events related to the treatments and the proportion of patients who discontinued the treatment because of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gisondi, MD, Principal Investigator — Universita di Verona
Locations (1):
- University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided